CLINICAL TRIAL: NCT01160926
Title: Dual Phase I Studies to Determine the Dose of Cediranib (AZD2171) or AZD6244 to Use With Conventional Rectal Chemoradiotherapy
Brief Title: Dual REctcal Angiogenesis or MEK Inhibition radioTHERAPY Trial
Acronym: DREAMtherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: 2 DLTs had been reported from first 4 patients on lowest possible dose cohort.
Sponsor: The Christie NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09_DOG03_184; 2009-016524-31 (EudraCT Number)
Record Dates: First submitted 2010-07-07; First posted 2010-07-13 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; capecitabine; radiotherapy; AZD6244; MEK inhibitor; AZD2171; Cediranib; VEGFR inhibitor; FLT-PET (fluoro-l-pyrimidine positron emission tomography); DCE-MRI (dynamic contrast enhanced magnetic resonance imaging)
MeSH Terms: conditions — Rectal Neoplasms | interventions — AZD 6244; cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD6244 + capecitabine + radiotherapy (Experimental): 10 days single-agent dosing AZD6244 Then 35 days dosing of AZD6244 in combination with standard chemoradiotherapy
  Interventions: Drug: AZD6244
- Cediranib + capecitabine + radiotherapy (Experimental): 10 days single agent dosing with Cediranib (AZD2171) then 35 days dosing of AZD2171 in combination with standard chemoradiotherapy
  Interventions: Drug: Cediranib (AZD2171)

INTERVENTIONS:
Drug: AZD6244 — Dose finding trial AZD6244 cohort 1 - 50mg bd AZD6244 cohort 2 - 75mg bd
  Capsule form, given for 10 days as single agent then for 35 days in combination with standard chemoradiotherapy
  Arms: AZD6244 + capecitabine + radiotherapy
Drug: Cediranib (AZD2171) — 10 days single agent dosing with Cediranib then 35 days in combination with standard chemoradiotherapy AZD2171 cohort 1 - 15mg od AZD2171 cohort 2 - 20mg od AZD2171 cohort 3 - 30mg od
  Oral tablets
  Other Names: AZD2171
  Arms: Cediranib + capecitabine + radiotherapy

SUMMARY:
To determine the maximum tolerated dose (MTD) of AZD6244 or AZD2171 when combined with pre-operative capecitabine and radiotherapy in patients with locally advanced rectal cancer.

DETAILED DESCRIPTION:
The best curative resection rates reported for patients with operable rectal cancer treated with standard chemoradiotherapy are approximately 50-60%.The pathological complete response rates are only 10-20%. Therefore, there is a need for more effective treatment. In this trial we will evaluate the combination of chemoradiotherapy with either a VEGFR (vascular endothelial growth factor receptor) or MEK (MAP Kinase)inhibitor.

Aims

1. Define the tolerability, MTD (maximum tolerated dose) and DLT (dose limiting toxicities) of chemoradiotherapy in combination with

   * cediranib, a VEGF receptor tyrosine kinase inhibitor that inhibits angiogenesis or
   * AZD6244, a potent MEK inhibitor that inhibits cell proliferation
2. Define a dose suitable for phase II evaluation
3. Test the impact of the combination on soluble and imaging (FLT-PET and DCEMRI/DWI) biomarkers to guide their use in phase II testing Summary Patients will receive standard chemoradiotherapy plus ascending doses of AZD6244 or cediranib from day -10 (relative to start of chemoradiotherapy) to day 35. If feasible, patients' tumours will be resected 10-12 weeks after treatment. Translational studies on available tissue and blood will be performed and DCE-MRI/DWI and FLT-PET will be carried out on 5 patients in the expanded cohort for AZD6244 (FLT-PET and DCE-MRI) and 5 patients in the expanded cohort for cediranib (DCE-MRI).

Cohorts Cediranib - 15mg od, 20mg od and 30mg od AZD6244 - 50mg bd and 75mg bd

ELIGIBILITY:
Inc Criteria:

* Histologically confirmed rectal adenocarcinoma
* MRI (magnetic resonance imaging) and triphasic CT (computerised tomography) defined locally advanced rectal cancer:

  * Mesorectal fascia involved or
  * Mesorectal fascia threatened or
  * Any T3 tumours < 5cm from the anal verge
* Primary resection unlikely to achieve clear margins
* No previous chemotherapy or radiotherapy for rectal cancer
* Bone marrow function: absolute neutrophil count ≥1.5 x109/l and platelet count >100 x109/l
* Hepatobiliary function: serum bilirubin <1.5 x upper limit of normal (ULN); serum ALP <5 x ULN; serum transaminase (AST or ALT) <2.5 x ULN
* Renal function: Serum creatinine clearance >50mL/min by either Cockcroft-Gault formula or EDTA (ethylenediaminetetraacetic acid) clearance
* ECOG PS(Eastern Cooperative Oncology Group Performance Status) 0-1
* Disease can be encompassed within a radical radiotherapy treatment volume
* No pre-existing condition which would deter radiotherapy, e.g. fistulas, severe ulcerative colitis, Crohn's disease, prior adhesions
* For women of child-bearing potential a negative pregnancy test is required and adequate contraceptive precautions such as a condom for their partner must be used. For men - adequate contraception must be used.
* Fit to receive all study treatments
* Able to comply with oral medication and protocol
* Signed, written and dated informed consent.
* Life expectancy ≥ 3 months.

Exc Criteria:

* Concurrent uncontrolled medical illness, or other previous/current malignant disease likely to interfere with protocol treatments
* Age<18
* Any pregnant, lactating women or potentially childbearing patients not using adequate contraception
* Previous chemotherapy or radiotherapy for rectal cancer
* Metastatic disease
* ECOG PS>1
* Patients who have very significant small bowel delineated within the radiation fields.
* Current or impending rectal obstruction (unless defunctioning stoma present), metallic colonic rectal stent in situ
* Pelvic sepsis.
* Uncontrolled cardiac, respiratory or other disease, or any serious medical or psychiatric disorder that would preclude trial therapy or informed consent.
* Cardiac conditions as follows:

  * Uncontrolled hypertension (resting BP ≥150/95mmHg despite optimal therapy)
  * Heart failure NYHA Class II or above
  * Prior or current cardiomyopathy
  * Atrial fibrillation with heart rate >100 bpm
  * Unstable ischaemic heart disease
* Refractory nausea and vomiting, chronic gastrointestinal diseases, or significant bowel resection that would preclude adequate absorption of trial drug
* Patients who are deemed unsuitable for surgery because of co-morbidity or coagulation problems.
* Recent (<14 days) major thoracic or abdominal surgery prior to entry into the study or a surgical incision that is not fully healed which would prevent administration of study treatment
* Known DPD (dihydropyrimidine dehydrogenase)deficiency
* Patients suffering from any condition that may affect the absorption of capecitabine or IMP (investigational medical product)
* Any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any patient known to have Hep B, Hep C or HIV
* Mean QTc with Bazetts correction >470msec in screening ECG or history of familial long QT syndrome

EXC CRITERIA (AZD6244 cohorts)

* KRAS (Kirsten ras sarcoma viral oncogene) wild-type
* Prior treatment with a MEK inhibitor
* Baseline LVEF (left ventricular ejection fraction) ≤50%

EXC CRITERIA (Cediranib cohorts)

* Known hypersensitivity to Cediranib or any of its excipients
* Greater than +1 proteinuria on two consecutive dipsticks taken no less than 1 week apart unless urinary protein < 1.5g in a 24 hr period or protein/creatinine ratio < 1.5.
* Significant haemorrhage (>30mL bleeding/episode in previous 3 months) or haemoptysis (>5mL fresh blood in previous 4 weeks)
* APTT ratio > 1.5 x ULN
* Arterial thromboembolic event (including ischemic attack) in the previous 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-07; Primary Completion 2013-10 (Actual); Study Completion 2016-11-04 (Actual)

PRIMARY OUTCOMES:
To determine the MTD (maximum tolerated dose) of AZD6244 or AZD2171 when combined with pre-operative capecitabine and radiotherapy in patients with locally advanced rectal cancer. | At point of surgery (10-12 weeks post treatment)

SECONDARY OUTCOMES:
Grade 3 or 4 toxicity | Up to point of surgery and long-term effects monitored for 3 years post treatment
Radiotherapy compliance | for the 5 weeks of chemoradiotherapy
MRI (Magnetic Resonance Imaging)Response Rate | 8 weeks post chemoradiation - at point of MRI scan
Histologically confirmed R0 resection rate | 10-12 weeks post chemoradiation - at time of surgery
Pathological Complete Response (pCR) | 10-12 weeks post chemoradiation - at point of surgery
Morbidity - post operative and long term | 3 years post chemoradiation
To explore biological and radiological markers of response or toxicity | Various timepoints up to point of surgery
  Tissue samples - from diagnostic sample, biopsy 6-8 days after single agent AZD6244/Cediranib and resection sample from surgery.
  Blood samples - screening, weeks 1, 3 and 5 during chemoradiotherapy and 8 weeks post chemoradiotherapy.
  FLT-PET scans - patients in AZD6244 cohorts only - at screening, after 10 days of dosing with single agent AZD6244 and 2 weeks post chemoradiation DCE-MRI scans - patients in both groups - at screening, after 10 days of dosing with single agent AZD6244/Cediranib and 2 weeks post chemoradiation

CONTACTS AND LOCATIONS:
Overall Officials: Mark P Saunders, MBBS, Principal Investigator — The Christie NHS Foundation Trust
Locations (1):
- The Christie NHS Foundation Trust, Manchester, United Kingdom